CLINICAL TRIAL: NCT05004012
Title: AnX/Ankon Navicam Magnetically Controlled Capsule Endoscopy Feasibility Study in Gastric Motility
Brief Title: Magnetically Controlled Capsule Endoscopy Feasibility Study in Gastric Motility
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lin Chang, MD, Principal Investigator, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB#20-001573
Record Dates: First submitted 2021-07-24; First posted 2021-08-13 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Gastroparesis; Dyspepsia
MeSH Terms: conditions — Gastroparesis; Dyspepsia | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: Four groups of participants will be studied: gastroparesis, functional dyspepsia, gastroparesis patients s/p G-POEM, and healthy controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Control (Other): No diagnosis of gastroparesis, functional dyspepsia, or prior G-POEM
  Interventions: Device: Magnetically Controlled Capsule Endoscopy
- Gastroparesis (Other): Patients with a diagnosis of gastroparesis meeting the inclusion criteria
  Interventions: Device: Magnetically Controlled Capsule Endoscopy
- Functional Dyspepsia (Other): Patients with a diagnosis of functional dyspepsia meeting the inclusion criteria
  Interventions: Device: Magnetically Controlled Capsule Endoscopy
- G-POEM (Other): Patients who received a G-POEM procedure meeting the inclusion criteria
  Interventions: Device: Magnetically Controlled Capsule Endoscopy

INTERVENTIONS:
Device: Magnetically Controlled Capsule Endoscopy — This is a diagnostic device for gastric disorders used to diagnose mucosal abnormalities. In this study it will be evaluated for use in gastric motility.

SUMMARY:
This is a feasibility study to assess the utility of magnetically controlled capsule endoscopy in the evaluation of gastroparesis and functional dyspepsia

DETAILED DESCRIPTION:
Gastroparesis and functional dyspepsia can both present with abdominal pain, dyspepsia, nausea, emesis, or early satiety. Gastroparesis is a syndrome defined as delayed gastric emptying. Functional dyspepsia is a symptom-based diagnosis in which the pathophysiology is multifactorial. Delayed gastric emptying is present in 25-35% of patients with functional dyspepsia. The study investigators propose the Navicam magnetically controlled capsule endoscopy (MCCE) system as a potential new method of evaluating gastric motility disorders. The MCCE is FDA approved for visualization of the stomach. The ability to visualize gastric peristalsis in real time, without interference from an endoscope, has never been demonstrated. The MCCE system could allow physicians to evaluate gastric motility with a test that has clear advantages over the current methods: it is fast, non-invasive, and has no radiation exposure, has artificial intelligence (AI) capabilities, while at the same time provides a visual assessment of the gastric anatomy. In this pilot feasibility study, the study investigators plan to enroll 5 male and female adult healthy volunteers, 5 male and female patients with gastroparesis, 5 male and female patients with functional dyspepsia (epigastric pain syndrome and/or postprandial distress syndrome with or without gastric emptying delay), and 2 patients with gastroparesis who have undergone a G-POEM procedure. The study investigators will compare gastric motor patterns in the different sections of the stomach and symptoms during fasting and a sham meal between groups.

ELIGIBILITY:
Inclusion Criteria

Must meet one of the following categories:

1. Gastroparesis

   Meets diagnostic criteria for gastroparesis:
   1. Evidence of delayed gastric emptying documented with a standard 2 hour or 4 hour gastric emptying scintigraphy exam
   2. Absence of mechanical obstruction
   3. Exhibits cardinal symptoms of early satiety, post-prandial fullness, nausea, vomiting, bloating, and upper abdominal pain

   Gastrointestinal cardinal symptom index (GCSI) score > 0 (i.e., the presence of at least mild severity of >1 of 3 symptoms of nausea/vomiting, postprandial fullness/early satiety, and/or bloating).
2. Functional Dyspepsia

   Meets Rome IV diagnostic criteria for functional dyspepsia:
   1. Criteria fulfilled for the last 3 months with symptom onset at least six months prior to diagnosis
   2. No evidence of organic, systemic, or metabolic disease that is likely to explain the symptoms on routine investigations (including at upper endoscopy)
   3. Meet criteria for Epigastric pain syndrome and/or Postprandial distress syndrome

   Epigastric Pain Syndrome At least 1 of the following symptoms at least 1 day per week
   1. Bothersome epigastric pain
   2. Bothersome epigastric burning

   Postprandial Distress Syndrome At least 1 of the following symptoms at least 3 days per week
   1. Bothersome postprandial fullness
   2. Bothersome early satiation
3. G-POEM

   1. The G-POEM procedure must have been performed at least 4 weeks prior to screening.
   2. GCSI score is < 3 which correlates to mild or less symptom severity.
4. Controls

None of the above conditions

Exclusion Criteria:

1. Another active disorder or treatment which could explain or contribute to symptoms in the opinion of the Investigator (including but not limited to gastric malignancy, neurological disorder, or heavy doses of strong anticholinergics).
2. Gastrectomy, fundoplication, vagotomy, bariatric surgery, post-surgical cause of gastroparesis, or gastric stimulation device surgically implanted within the last year. Prior G-POEM procedure for gastroparesis is allowed for the group of post-G-POEM study subjects.
3. Dysphagia, swallowing disorder
4. Suspected bowel obstruction or perforation
5. Gastric or parenteral feeding within 4 weeks of screening
6. Pregnancy or nursing
7. History of an eating disorder within 2 years of screening
8. Recent history (within six months of screening) of Alcohol Use Disorder or Substance Use Disorder as defined in DSM-5.
9. Uncontrolled thyroid disease
10. Unstable cardiac, respiratory, hepatic or renal disease
11. Evidence of uncontrolled blood glucose (including HbA1C >9 or metabolic crisis in past 60 days).
12. Use of prohibited medication or medication with anti-nausea, antiemetic, neuromodulating, or prokinetic effect within 2 weeks of the screening visit EXCEPT when administered on a stable daily dosing schedule (stable for at least 1 month prior to the screening visit).
13. Use of as needed or daily opioids within the past 1 month.
14. Pyloric injection of neurotoxins (e.g. botulinum type A or B) within 3 months of the Screening visit.
15. Altered mental status (e.g., hepatic encephalopathy) that limits the ability to swallow a capsule
16. Expected to have Magnetic Resonance Imaging (MRI) examination within 30 days.
17. No reliable contact information - no phone, no permanent address.
18. Pacemaker or ICD
19. Inability to avoid using the bathroom for urination and/or bowel movements for the duration of the study.
20. Metal Implant (ie metal hip arthroplasty, surgical mesh, coronary or arterial stent)
21. Prior bowel surgery
22. Severe claustrophobia
23. Any other reason as determined by the Investigator which may lead to an unfavorable risk-benefit of study participation, may interfere with study compliance, or may confound study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Frequency and direction of contractions | Through study completion, an average of 1 year
  Physiologic parameter measuring the frequency and direction of stomach contractions
Number and location of luminal transit markers in the antrum, fundus, and overall | Through study completion, an average of 1 year
  Physiologic parameter measuring the number and location of luminal transit markers in the stomach
Largest diameter of the pylorus | Through study completion, an average of 1 year
  Physiologic parameter measuring the diameter of the pylorus
Dyspepsia Severity Scale symptom ratings at baseline and during the study at timepoints with discomfort if present. | Through study completion, an average of 1 year
  Evaluating the dyspepsia Severity Scale symptom ratings (range of score 0-20) at baseline and during the study at timepoints with discomfort if present.
Procedure related adverse events | Through study completion, an average of 1 year
  Procedure related adverse events during or after the study session

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chang, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacy BE, Talley NJ, Locke GR 3rd, Bouras EP, DiBaise JK, El-Serag HB, Abraham BP, Howden CW, Moayyedi P, Prather C. Review article: current treatment options and management of functional dyspepsia. Aliment Pharmacol Ther. 2012 Jul;36(1):3-15. doi: 10.1111/j.1365-2036.2012.05128.x. Epub 2012 May 16. PMID 22591037
- [Background] Camilleri M, Parkman HP, Shafi MA, Abell TL, Gerson L; American College of Gastroenterology. Clinical guideline: management of gastroparesis. Am J Gastroenterol. 2013 Jan;108(1):18-37; quiz 38. doi: 10.1038/ajg.2012.373. Epub 2012 Nov 13. PMID 23147521
- [Background] Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Development and validation of a patient-assessed gastroparesis symptom severity measure: the Gastroparesis Cardinal Symptom Index. Aliment Pharmacol Ther. 2003 Jul 1;18(1):141-50. doi: 10.1046/j.1365-2036.2003.01612.x. PMID 12848636
- [Background] Revicki DA, Rentz AM, Tack J, Stanghellini V, Talley NJ, Kahrilas P, De La Loge C, Trudeau E, Dubois D. Responsiveness and interpretation of a symptom severity index specific to upper gastrointestinal disorders. Clin Gastroenterol Hepatol. 2004 Sep;2(9):769-77. doi: 10.1016/s1542-3565(04)00348-9. PMID 15354277
- [Background] Carbone F, Vanuytsel T, Tack J. Analysis of Postprandial Symptom Patterns in Subgroups of Patients With Rome III or Rome IV Functional Dyspepsia. Clin Gastroenterol Hepatol. 2020 Apr;18(4):838-846.e3. doi: 10.1016/j.cgh.2019.07.053. Epub 2019 Aug 5. PMID 31394286